CLINICAL TRIAL: NCT01839136
Title: Gametes Transfer vs. Embryo Transfer for Women Undergoing Assisted Reproductive Techniques: a Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low pregnancy rates in both groups
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Wellington P Martins, MD, Physician and researcher, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 03332812.0.0000.5440
Record Dates: First submitted 2013-04-21; First posted 2013-04-24 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Infertility
Keywords: Assisted Reproductive Techniques; Health Services Accessibility; Ovulation Induction; Embryo Transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrauterine transfer of gametes (Experimental): After the oocyte retrieval, the oocytes will be selected depending on the morphology of the granular cells. The transfer will be conducted in up to 2 hours after the oocytes collection, when the semen and up to 3 oocytes will be transferred. Surplus oocytes will be cryopreserved for future use. We will use a Sydney catheter (Cook Medical Inc., Bloomington, IN, USA) coupled to a 1 mL syringe to perform the transfer. The catheter will be loaded with oocytes and semen prepared in the following sequence: 10 µL of the prepared semen, a small space of air, 20 µL of the medium containing the oocytes, another small space of air and more 10 µL of prepared semen. The catheter will be placed through the endocervical canal up to the endometrial cavity guided by transabdominal ultrasound, where the liquid will be released. We will try to place the point of the catheter 1.0-1.5cm before touching the fundus of the endometrial cavity and release the liquid slowly, in approximately 30 seconds.
  Interventions: Procedure: Intrauterine transfer of gametes
- intrauterine transfer of embryos (Active Comparator): The oocytes will be denuded and those considered to be mature will be selected for fertilization up to the number of seven. In vitro fertilization will be performed and up to two embryos will be transferred 2-3 days after the oocyte retrieval. The other embryos will be cryopreserved for future use. We will use Sidney catheter (Cook Medical Inc.) coupled to a 1 mL syringe to perform the transfer. The catheter will be loaded with embryos in the following sequence: 10 µL of culture medium, a small space of air, 20 µL of the medium containing embryos, another small space of air, and more 10 µL of culture medium. The catheter will be placed through the endocervical canal up to the endometrial cavity, guided by transabdominal ultrasound, where the liquid will be released. We will try to place the point of the catheter 1.0-1.5cm before touching the fundus of the endometrial cavity and release the liquid slowly, in approximately 30 seconds.
  Interventions: Procedure: Intrauterine transfer of embryos

INTERVENTIONS:
Procedure: Intrauterine transfer of gametes
  Arms: Intrauterine transfer of gametes
Procedure: Intrauterine transfer of embryos
  Arms: intrauterine transfer of embryos

SUMMARY:
Background: The cost for the treatment of infertility are limiting for the health care access, particularly if we consider that the success rate per cycle is approximately 35%. Alternative regimens for controlled ovarian stimulation (COS)have been described in the medical literature, that lead to a lower cost, fewer injections and less risk of adverse events, particularly ovarian hyperstimulation syndrome. Furthermore, some services report excellent results with less manipulation as possible, which reduces the cost of laboratory of human and ethically be considered less complicated once fertilization occurs in the uterus and not in vitro.

Objectives: The main objective is to compare the reproductive outcomes between intrauterine transfer of gametes (TG) and embryos (TE), the secondary objective is to estimate the average number of eggs that are raised when using an EOC reduced cost.

Methods: This study will be conducted in the area of Human Reproduction, Department of Gynecology and Obstetrics Hospital of the FMRP-USP. We will conduct an open controlled study with random allocation of the participants in a 1:1 ratio, and we plan to include 100 participants. All participants will undergo an EOC reduced cost. We will compare the chance of the treatment (TE or TG) result in a live birth and clinical pregnancy per woman allocated and to estimate the number of oocytes retrieved considering all participants.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing ART requiring COS, oocyte retrieval and embryo transfer at the fertility clinic of the university Hospital of the Medical School of Ribeirao Preto, University of Sao Paulo, Brazil.
* Age = 18-40 years
* BMI = 18-30 Kg/m²
* Antral follicle count (AFC) ≥ 5
* Semen concentration and progressive motility above the percentile 2.5 of the fertile men (Cooper et al. 2010): sperm concentration > 9X 10⁶/mL, and progressive motility > 28%.

Exclusion Criteria:

* None

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Live birth | 9 months

SECONDARY OUTCOMES:
Clinical pregnancy | 2 months
Number of oocytes retrieved | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Setor de Reproducao Humana do HC-FMRP-USP, Ribeirão Preto, São Paulo, Brazil